CLINICAL TRIAL: NCT06021769
Title: Longitudinal Assessment of Pessary Experience
Brief Title: Pessary Experience Study
Status: Recruiting | Type: Observational
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Monique Vaughan, MD, Assistant Professor, University of Virginia
Other Study IDs: HSR220160
Record Dates: First submitted 2023-08-26; First posted 2023-09-01 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Pelvic Organ Prolapse; Stress Urinary Incontinence
Keywords: pessary
MeSH Terms: conditions — Pelvic Organ Prolapse; Urinary Incontinence, Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Women being fitted with pessaries: Women being fitted with pessaries as standard of care will be eligible to participate. They will be asked to complete a recorded verbal interview and written questionnaires the day they have their pessaries fitted and at their follow-up clinic appointments at 4-6 weeks, 3 months, 6 months, and 12 months. Another recorded video interview will be completed at the 12 month appointment.
  Interventions: Other: Observational only

INTERVENTIONS:
Other: Observational only — No intervention

SUMMARY:
Pessaries are silicone devices inserted into the vagina for treatment of pelvic organ prolapse or stress urinary incontinence. They are adequate treatment options for patients who are poor surgical candidates, those who decline surgical intervention, or as a temporizing measure in those ultimately planning surgery. Most studies suggest that about 75% of patients are able to be successfully fit with a pessary, but about 50% discontinue pessary use within 12 months of initiation. The purpose of this study is to determine why pessaries are discontinued.

DETAILED DESCRIPTION:
Pessaries are silicone devices inserted into the vagina for treatment of pelvic organ prolapse or stress urinary incontinence. They are adequate treatment options for patients who are poor surgical candidates, those who decline surgical intervention, or as a temporizing measure in those ultimately planning surgery. Most studies suggest that about 75% of patients are able to be successfully fit with a pessary, but about 50% discontinue pessary use within 12 months of initiation.

Research concerning pessary discontinuation is currently focused on identifying factors that will predict outcomes of pessary use. It is generally agreed upon that pessaries are one of the favored option to conservatively treat pelvic organ prolapse or stress urinary incontinence, but there is not sufficient consensus on the rate of discontinuation, factors leading to discontinuation, and patient satisfaction.

Most studies recorded reasons for discontinuation and any adverse events. Patients' reasons for discontinuation of pessary use included frequent expulsion, difficulty removing pessary, new or worsening urinary incontinence, vaginal erosion, and pain/discomfort. Significant side effects or adverse events included vaginal discharge and erosion.

Several studies focused on anatomic and medical variables that were correlated to pessary discontinuation. A univariate analysis of factors contributing to discontinuation conducted by Yimphong et al.1 found that higher BMI and history of pelvic surgery were significant in predicting discontinuation. Similarly, Panman2 et al. conducted a multivariate analysis that found higher BMI was a significant factor. Panman et al. also found that both younger age and weaker pelvic floor muscles were predictors for discontinuation. The former finding is further supported by Umchanger et al., which cited that 33% of patients who discontinued pessary use within three months were generally less than 65 years. Umchanger et al. hypothesized that despite data suggesting that pessaries are as effective as surgery, younger patients may maintain the misconception that pessaries are not as effective.

Despite the data suggesting contributing factors such as BMI and age, none of the reviewed studies captured the qualitative reasoning behind patients' decisions. Only a few of the studies investigate patients' satisfaction with pessary use, quality of life, or opinion on their treatment.

Pessary use has been correlated to a wide variety of factors, such as a patient's medical history, anatomic characteristics, beliefs about pessary use, and personal satisfaction with treatment. Based on this review, a qualitative analysis of patient experience and priorities as they decide to continue or discontinue pessary use would be incredibly helpful for counseling and educating future patients when they are making treatment decisions about pessaries.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking women aged 18 years or older
* Choosing to undergo a pessary fitting for symptomatic pelvic organ prolapse and/or stress urinary incontinence at the University of Virginia Pelvic Medicine and Reconstructive Surgery clinic
* Willingness and ability to comply with scheduled visits and study procedures.
* Successful pessary fitting

Exclusion Criteria:

* Pregnant women
* Prisoners
* Cognitively impaired
* Non-English speaking subjects
* Patients who cannot comply with pessary check visits
* Active vaginal infection
* Vaginal malignancy
* Genitourinary tract fistula

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women in the area surrounding the University of Virginia who have stress urinary incontinences or pelvic organ prolapse.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-06-12 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Qualitative analysis | up to 1 year after pessary fitting
  Perform a patient-centered, qualitative analysis of pessary discontinuation
Pelvic Floor symptom improvement as related to quality of life | up to 1 year after pessary fitting
  Assess changes in pelvic floor symptoms and quality of life before and after pessary use as measured by validated questionnaires
Discontinuation of pessaries | up to 1 year after pessary fitting
  Rates of discontinuation at 1 year
Why do women discontinue using pessaries? | up to 1 year after pessary fitting
  Factors significantly associated with discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Monique Vaughan, MD, Principal Investigator — Assistant Professor
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yimphong T, Temtanakitpaisan T, Buppasiri P, Chongsomchai C, Kanchaiyaphum S. Discontinuation rate and adverse events after 1 year of vaginal pessary use in women with pelvic organ prolapse. Int Urogynecol J. 2018 Aug;29(8):1123-1128. doi: 10.1007/s00192-017-3445-x. Epub 2017 Aug 16. PMID 28815277
- [Background] Panman CM, Wiegersma M, Kollen BJ, Burger H, Berger MY, Dekker JH. Predictors of unsuccessful pessary fitting in women with prolapse: a cross-sectional study in general practice. Int Urogynecol J. 2017 Feb;28(2):307-313. doi: 10.1007/s00192-016-3107-4. Epub 2016 Aug 15. PMID 27525693
- [Background] Umachanger JK, Marcussen ML, Boggild H, Kjaergaard N, Glavind K. First-line treatment of pelvic organ prolapse and discontinuation of pessary treatment. Int Urogynecol J. 2020 Sep;31(9):1813-1819. doi: 10.1007/s00192-020-04338-w. Epub 2020 May 24. PMID 32447418